CLINICAL TRIAL: NCT06009263
Title: Effect of Open Chain Versus Closed Chain Segmental Control Exercises on Cross Sectional Area of Lumbar Multifidus Muscle in Chronic Mechanical Low Back Pain
Brief Title: Effect of Open Chain Versus Closed Chain Segmental Control Exercises on CSA of Lumbar Multifidus Muscle in Chronic MLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haytham M Elhafez, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/007/002763
Record Dates: First submitted 2023-08-13; First posted 2023-08-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Mechanical Low Back Pain
Keywords: Mechanical LBP; Cross Sectional Area; Multifidus muscle
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Group will receive ultrasound and TENS as conventional treatment
Who Masked: Participant
Masking Description: Group will receive open chain segmental control exercises versus closed chain segmental control exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Sham Comparator): The participants will receive conventional treatment in the form of TENS and Ultrasound.
  Interventions: Other: Conventional treatment
- Intervention 1 (Experimental): The participants will receive "open chain segmental control exercises" plus conventional treatment in the form of TENS and Ultrasound.
  Interventions: Other: Open chain segmental control
- Intervention 2 (Experimental): The participants will receive "closed chain segmental control exercises" plus conventional treatment in the form of TENS and Ultrasound.
  Interventions: Other: Closed chain segmental control

INTERVENTIONS:
Other: Conventional treatment — Application of ultrasound and transcutaneous electrical nerve stimulation "TENS" for mechanical low back pain.
  Arms: Control
Other: Open chain segmental control — Application of "open chain segmental control exercises" As well as, application of ultrasound and transcutaneous electrical nerve stimulation "TENS" for mechanical low back pain.
  Arms: Intervention 1
Other: Closed chain segmental control — Application of "closed chain segmental control exercises" As well as, application of ultrasound and transcutaneous electrical nerve stimulation "TENS" for mechanical low back pain.
  Arms: Intervention 2

SUMMARY:
To investigate the effect of adding open versus closed chain segmental control exercises to conventional treatment program on pain intensity, lumbar ROM, and CSA of multifidus muscle.

DETAILED DESCRIPTION:
* To investigate the effect of adding open versus closed chain segmental control exercises to conventional treatment program on pain intensity.
* To investigate the effect of adding open versus closed chain segmental control exercises to conventional treatment program on lumber ROM.
* To investigate the effect of adding open versus closed chain segmental control exercises to conventional treatment program on CSA of multifidus muscle.
* To investigate the effect of adding open versus closed chain segmental control exercises to conventional treatment program on lumber function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic low back pain from both genders their age will be ranged and divided into three groups from 25-55 years.
2. Participants with chronic low back pain lasting for more than 6 Months.
3. A patient who can follow the command.
4. A patient who can do exercise.

Exclusion Criteria:

1. Low back pain patients with a history of severe neurological disease or orthopedic disease.
2. History of Psychological Disorder.
3. Unhealthy Patient.
4. Pregnant women.
5. Patient with a spinal tumor.
6. History of any operation related to spine. Ex. Vertebral fracture or dislocation.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cross sectional area of multifidus muscle | Pre and Post measurement (12 weeks)
  Cross sectional area of multifidus muscle
Pain intensity | Pre and Post measurement (12 weeks)
  Measured by VAS (from 0 to 10; 0 means no pain and 10 means worst pain)

SECONDARY OUTCOMES:
ROM of lumbar spine | Pre and Post measurement (12 weeks)
  Measuring ROM of lumbar spine
Functional ability of lumbar spine | Pre and Post measurement (12 weeks)
  Questionnaire for measuring lumbar activities (lower score means better and higher score means worse)

CONTACTS AND LOCATIONS:
Overall Officials: Haytham M Elhafez, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No